CLINICAL TRIAL: NCT03190954
Title: Brain Dopaminergic Signaling in Opioid Use Disorders (OUD)
Brief Title: Brain Dopaminergic Signaling in Opioid Use Disorders
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 170114; 17-AA-0114
Record Dates: First submitted 2017-06-16; First posted 2017-06-19 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01-12

CONDITIONS: Normal Physiology; Opioid Use Disorders
Keywords: Raclopride; NNC-112; Functional Magnetic Resonance Imaging (fMRI); Dopamine D1 Receptor; D2 Receptors
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- [11C]NNC-112 (Placebo Comparator): [11C]NNC-112 PET scan obtained without any drug intervention to measure dopamine D1 receptors. Blind N/A
  Interventions: Drug: [11C]NNC-112
- [11C]raclopride plus drug (Active Comparator): Methylphenidate 60 mg. po will be given 60 minutes prior to [11C]raclopride scan to measure striatal dopamine release. MRI scan to follow end of PET scan. Subject blind as to drug administration.
  Interventions: Drug: [11C]raclopride plus drug; Drug: [11C]NNC-112
- [11C]raclopride plus placebo (Placebo Comparator): Placebo (po) will be given 60 minutes prior to [11C]raclopride scan to measure baseline dopamine D2 receptors. MRI scan to follow end of PET scan. Subject blind as to drug administration.
  Interventions: Drug: [11C]raclopride plus placebo; Drug: [11C]NNC-112

INTERVENTIONS:
Drug: [11C]raclopride plus placebo — Placebo (po) will be given 60 minutes prior to [11C]raclopride scan to measure baseline dopamine D2 receptors. MRI scan to follow end of PET scan. Subject blind as to drug administration.
  Arms: [11C]raclopride plus placebo
Drug: [11C]raclopride plus drug — Methylphenidate 60 mg. po will be given 60 minutes prior to [11C]raclopride scan to measure striatal dopamine release. MRI scan to follow end of PET scan. Subject blind as to drug administration.
  Arms: [11C]raclopride plus drug
Drug: [11C]NNC-112 — [11C]NNC-112 PET scan obtained without any drug intervention to measure dopamine D1 receptors. Blind N/A

SUMMARY:
Background:

The chemical messenger dopamine carries signals between brain cells. It may affect addiction. Heavy use of pain medicines called opioids may decrease the amount of dopamine available to the brain. Researchers want to study if decreased dopamine decreases self-control and increases impulsiveness.

Objective:

To learn more about how opiate use disorder affects dopamine in the brain.

Eligibility:

Adults 18-80 years old who are moderate or severe opiate users

Healthy volunteers the same age

Design:

Participants will first be screened under another protocol. They will:

* Have a physical exam
* Answer questions about their medical, psychiatric, and alcohol and drug use history
* Take an MRI screening questionnaire
* Give blood and urine samples
* Have their breath tested for alcohol

Participants will have up to 3 study visits.

They will have 2-3 positron emission tomography (PET) scans. A radioactive chemical will be injected for the scans. Participants will lie on a bed that slides in and out of the donut-shaped scanner. A cap or plastic mask may be placed on the head.

Vital signs will be taken before and after the PET scans.

Participants will get capsules of placebo or the study drug. They will rate how they feel before, during and after.

Participants will have their breath and urine tested each day.

Participants will have magnetic resonance imaging (MRI) scans. They will lie on a table that slides into a cylinder in a strong magnetic field. They may do tasks on a computer screen while inside the scanner.

Participants will have tests of memory, attention, and thinking.

Participants will wear an activity monitor for one week....

DETAILED DESCRIPTION:
Objectives: Primary objective is to assess whether the balance between dopamine D1 (D1R) and D2 receptors (D2R) signaling in striatum is disrupted in participants with an opioid use disorder (OUD) who are on opioid agonist medication (MAT+: methadone or buprenorphine) relative to OUD participants treated with the opioid antagonist medication naltrexone and OUD participants in recovery and not being treated with medications (MAT-). Secondary objectives are to assess how striatal D1R to D2R availability (assessed with PET) influences: (1) striatal dopamine (DA) release; (2) the function of brain reward and self-control networks (assessed with task fMRI activation and with resting functional connectivity, RFC) and (3) behavior (locomotor activity and neuropsychological tests); (4) to assess if DA increases, as induced by oral methylphenidate (MP), improve the function of brain reward and control networks in OUD; and (5) to assess if there is recovery after protracted treatment (comparing treated and non-treated) by repeating fMRI at 6 month follow-up.

Study population: We will complete studies in 180 (n=180) subjects: N=60 healthy control adults and N=120 OUD participants (60 MAT+, 30 naltrexone-treated and 30 MAT-) aged 18-80 (male/female) will be included.

Design: Single-blind. Participants will undergo three scans with positron emission tomography (PET): one with [11C]NNC-112 to assess baseline D1R, another with [11C]raclopride after placebo to assess baseline D2R and a third one with [11C]raclopride after MP administration (60mg oral) to assess striatal DA release (assessed as the difference in specific binding of [11C]raclopride between baseline and MP). In addition, participants will undergo two imaging sessions with MRI to assess functional reactivity to drug-cues and to a measure of self-control (delayed discounting task), to assess RFC and to obtain structural brain measures (including diffusion tensor imaging, DTI). One of the sessions will be done under baseline conditions (no drug administered) and the other after MP (about one hour after the [11C]raclopride MP scan is completed). Neuropsychological tests (NP) and accelerometers will be used to assess cognitive performance and locomotor activity respectively.

Outcome Measures: Main outcome: (1) Differences in D1R to D2R striatal ratio between participants with an OUD and controls and between MAT+, naltrexone, and MAT- groups. Secondary outcomes: Correlations between striatal D1R to D2R and (1) striatal DA release; (2) fMRI activation in reward and controls networks (assessed with cue-reactivity and delay discounting tasks, and with RFC) and (3) NP performance and locomotor activity. (4) Differences in fMRI activation and RFC after MP when compared with baseline measures.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy Volunteer Participants

1. Males or females between 18 and 80 years of age.
2. Ability to provide written informed consent.

MAT- Opiate Use Disorder (OUD) Participants

1. Males or females between 18 and 80 years of age.
2. Ability to provide written informed consent.
3. DSM-5 diagnosis of a moderate or severe OUD (established through history and clinical exam).
4. Minimum of 3 months since last regular use of opioids (no more than 1x/week in the past 3 months as assessed by self-report).
5. Minimum 3 year history of past opiate abuse - self-report.
6. Must have consumed opiates at least 5 days per week (past opioid use) as per self-report.
7. Currently not receiving medications for OUD and a minimum of 3 months since last regularly taking medications for OUD (methadone, buprenorphine or naltrexone) as per self-report.

MAT+ OUD Participants

1. Males or females between 18 and 80 years of age.
2. Ability to provide written informed consent.
3. DSM-5 diagnosis of a moderate or severe OUD (established through history and clinical exam).
4. Active or non-active abuse of opiates.
5. Minimum 3 year history of opiate abuse as per self-report.
6. Must have consumed at least 5 days per week (prior opiate use) as per self-report.
7. Receiving opioid agonist therapy for OUD (e.g., methadone or buprenorphine) and must have taken for at least one week before imaging study

Naltrexone OUD Participants

1. Males or females between 18 and 80 years of age.
2. Ability to provide written informed consent.
3. DSM-5 diagnosis of a moderate or severe OUD (established through history and clinical exam).
4. Active or non-active abuse of opiates.
5. Minimum 3 year history of opiate abuse as per self-report.
6. Must have consumed at least 5 days per week (prior opiate use) as per self-report.
7. Receiving naltrexone treatment for their OUD and must have taken at least one week before imaging study.

For all groups of subjects regarding inclusions 1 & 2:

* 1: OUD and HV subjects who are age 66-80 may be included in this study except they will not receive the methylphenidate and subsequent PET/[11C]raclopride and MRI scans. They will receive the placebo (Phase D) and subsequent PET/[11C]raclopride and MRI scans.
* 2: Source documentation for the subject s ability to provide written informed consent will be a note in CRIS documenting that the subject is alert and oriented to person, place, and time; and/or an unremarkable neurological examination; dated on or before the date of consent.

EXCLUSION CRITERIA:

Healthy Volunteer Subjects

1. Current DSM-5 diagnosis of a psychiatric disorder (other than nicotine/caffeine use) that requires/required daily psychoactive medications (antidepressant, antipsychotics, stimulants, benzodiazepines or barbiturates) in the past two months and that could impact brain function at the time of the study as determined by history and clinical exam.
2. The following current chronically used (2 months) medications are exclusionary: stimulant or stimulant-like medications (amphetamine, methylphenidate, modafinil); opioid analgesics; antianginal agents; antiarrhythmics; systemic corticosteroids; anticholinergics; anticoagulants; anticonvulsants; antidepressants; antihistamines (sedating); beta-blocker antihypertensives; antineoplastics; antiobesity; antipsychotics; anxiolytics (benzodiazepine or barbiturates); lithium; muscle relaxants; psychotropic drugs not otherwise specified (nos); sedatives/hypnotics, systemic steroids. Note that nicotine and/or caffeine is not exclusionary. Subjects on stable antihypertensive medications (except for beta blockers) may be included provided they are on a clinically stable dose for at least a month [BP must be <= 140/90 if participating in MP or placebo administration scans (Phases A &B); or BP must be <= 160/100 if participating in placebo administration scan (Phase D)].
3. Current continuous treatment (> 3 weeks) with methadone, buprenorphine or naltrexone.
4. Current major medical problems that can permanently impact brain function (e.g., CNS: including seizures, psychosis, stroke, severe depression, Alzheimer s, Parkinson s disease, Traumatic brain injury; Cardiovascular: including uncontrolled hypertension [BP > 140/90] and clinically significant EKG results except bradycardia; and HIV+) as determined by history.
5. Clinically significant laboratory findings that could impact brain function or study procedures (e.g., active infections, significant EKG results, hepatic or renal failure) will be exclusionary.
6. Have had previous radiation exposure (from X-rays, PET scans, or other exposure) that, with the exposure from this study, would exceed NIH annual research limits as determined by medical history and physical exam.
7. Head trauma with loss of consciousness for more than 30 minutes as determined by medical history and physical exam.
8. Pregnant and/or currently breast-feeding. Females of childbearing potential (age 60 or less) will undergo a urine pregnancy test that must be negative to participate. Urine pregnancy tests will be repeated on subsequent days of study.
9. Presence of ferromagnetic objects in the body that are contraindicated for MRI (pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips, metallic prostheses, permanent eyeliner, implanted delivery pump, or shrapnel fragments) or fear of enclosed spaces - self-report checklist.
10. Personal or family history (parents or siblings) for cerebral aneurysm.
11. Past or present history of chest pain and trouble breathing with activity.
12. Glaucoma as assessed by medical history.
13. Cannot lie comfortably flat on their backs for up to 2 hours in the PET and MRI scanners self-report.
14. Weight > 400 pounds, which is the maximum weight the PET scanner can hold.
15. Study investigators and staff, as well as their superiors, subordinates and immediate family members (adult children, spouses, parents, siblings).
16. *Non-English speakers (must also be able to read and comprehend English).

OUD Subjects

1. DSM-5 diagnosis of a psychiatric disorder that requires daily use of antipsychotic medications (schizophrenia or any other psychotic disorder) at the time of the study as determined by history and clinical exam.
2. Currently on antipsychotic medications. Subjects on stable antihypertensive medications may be included provided they are clinically stable [BP must be <= 140/90 if participating in MP administration scan (Phases A & B); or BP must be <= 160/100 if participating in placebo administration scan (Phase D). OUD subjects who are taking a stimulant medication may participate in the study, except that they will be asked to not take their prescribed stimulant medication on the days of the [11C]raclopride scans.
3. Current continuous treatment (> 3 weeks) with methadone or buprenorphine for MAT- OUD participants; or naltrexone for MAT+ OUD participants; or agonist treatment (methadone or buprenorphine) for OUD participants treated with Naltrexone.
4. Current major medical problems that can permanently impact brain function (e.g., CNS: including seizures, psychosis, stroke, severe depression, Alzheimer's, Parkinson s disease, Traumatic brain injury; Cardiovascular: including uncontrolled hypertension [BP > 140/90 excludes from participating in MP administration scan (Phases A & B); or BP > 160/100 excludes from participating in placebo administration scan (Phase D)] and clinically significant EKG results except bradycardia; and HIV+) as determined by history. However, OUD subjects who have hypertension and/or certain non-significant EKG results may still be included in this study except they will not receive the methylphenidate and subsequent PET/RAC and/or MRI scans, but will receive the placebo and subsequent PET/RAC and/or MRI scans as long as their BP's are <= 160/100 based on BP's obtained during initial H&P.
5. Clinically significant laboratory findings that could impact brain function or study procedures (e.g., active infections, significant EKG results, hepatic or renal failure) will be exclusionary.
6. Have had previous radiation exposure (from X-rays, PET scans, or other exposure) that, with the exposure from this study, would exceed NIH annual research limits as determined by medical history and physical exam.
7. Head trauma with loss of consciousness for more than 30 minutes as determined by medical history and physical exam.
8. Pregnant and/or currently breast-feeding. Females of childbearing potential (age 60 or less) will undergo a urine pregnancy test that must be negative to participate. Urine pregnancy tests will be repeated on subsequent days of study.
9. Presence of ferromagnetic objects in the body that are contraindicated for MRI (pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips, metallic prostheses, permanent eyeliner, implanted delivery pump, or shrapnel fragments) or fear of enclosed spaces - self-report checklist. However, OUD subjects who are contraindicated for MRI participation, or the study team cannot access prior surgical records to confirm that a subject is cleared for MRI, may still participate in all aspects of the study except MRI. If it is discovered during the clinical brain MRI or after enrollment onto the study that the subject experiences anxiety or becomes claustrophobic, we will discontinue the MRI portion of the study and he/she can continue to participate in all other aspects of the study.
10. Personal or family history (parents or siblings) for cerebral aneurysm. Participant may be included in the PL administration with PET/RAC and/or MR but is excluded from the MP administration and subsequent PET/RAC and/or MR scan if history is reported.
11. Past or present history of chest pain and trouble breathing with activity. Participant may be included in the PL administration with PET/RAC and/or MR but is excluded from MP administration and subsequent PET/RAC and/or MR scan if history is reported.
12. Glaucoma as assessed by medical history. Participant may be included in the PL administration with PET/RAC and/or MR but is excluded from MP administration and subsequent PET/RAC and/or MR scan if history of glaucoma reported.
13. Cannot lie comfortably flat on their backs for up to 2 hours in the PET and MRI scanners self-report.
14. Weight > 400 pounds, which is the maximum weight the PET scanner can hold.
15. Study investigators and staff, as well as their superiors, subordinates and immediate family members (adult children, spouses, parents, siblings).
16. *Non-English speakers (must also be able to read and comprehend English).

    Additional exclusion criteria for MAT+ / MAT- / Naltrexone OUD participants:
17. Participation in a court ordered residential treatment program.

Note that subjects will not be excluded from enrollment onto this study if their urine test or breath alcohol level (BAL) is positive for drugs/alcohol on initial screening. The following guidelines will be followed for positive drug/alcohol screens on study procedure days:

If a Healthy Volunteer subject s urine drug screen test or breath alcohol (>0.08%) is positive on days involving imaging (MRI and/or PET) and NP testing, the procedures will be postponed and rescheduled. We will allow for up to 3 rescheduled study days resulting from positive urine drug/breath alcohol screens. If urine drug screen is positive for THCCOOH only, a saliva drug screen will be performed and subject may proceed with study day testing procedures if saliva results for THC are negative. If we are unable to perform the saliva drug screen in HV s for any reason, the study day procedures will be postponed. If the urine/saliva drug test is positive on the third rescheduled visit, the participant will be withdrawn from the study. Saliva THC is not required for determining eligibility.

If an OUD subject s urine drug screen test or breath alcohol (>0.08%) is positive for drugs the procedures will not be postponed. If urine drug screen is positive for THC-COOH, a saliva drug screen will be performed to verify if THC is present. If we are unable to perform the

saliva drug screen for any reason, the subject may still participate in the study on the same day. Positive results for drugs other than opiates will be considered at the time of data analysis as a co-variate. Saliva THC is not required for determining eligibility.

*The intent of the research has no prospect of direct benefit to the subject. Therefore, we are excluding non-English speakers in this research study since it includes the administration of questionnaires, surveys and assessments that are validated for English, although some are available in Spanish. In addition, our fMRI paradigms (particularly the Delay Discounting task) require that the subject be able to speak, read and comprehend English.

For exclusion #2 in the healthy volunteers and the OUD groups, subjects on stable antihypertensive medications may be included provided they are on a clinically stable dose for at least a month with BP s on initial screening obtained under the 14AA0181 protocol are <= 140/90 if participating in MP administration scans (Phases A & B). If these subject groups are not taking antihypertensive medications, they will receive the placebo (Phase D) provided that BP s on initial screening obtained under the 14AA0181 protocol are <= 160/100.

Abnormal lab results will be reviewed by a clinician for a determination of whether results are not clinically significant (NCS) for inclusion on the study. For example, if an OUD subject has a positive Hep C antibody with or without a detected viral load, we will not exclude solely based on abnormal lab results since many OUD subjects have prior exposure to Hep C and up to 25% of exposed subjects have spontaneous clearance of the virus. Rather, we will evaluate the abnormal lab results on an individual basis to determine whether subject can proceed with the study. The subject will be counseled to follow up with their PCP for management.

Also, note that at any time during participation in this study if any subject expresses that he/she wants to get treatment for their OUD, we will immediately refer him/her to a treatment program. If the subject was enrolled as a participant in recovery (MAT-), the subject will be withdrawn from the study at that time. No OUD medications will be stopped or held for participation in this protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
Differences in D1R to D2R striatal ratio and in DA release between participants with an OUD and controls and between MAT+, naltrexone, and MAT- groups. | End of study
  To assess whether the balance between D1R and D2R in striatum and in DA release is disrupted in participants with an opioid use disorder (OUD) who are being treated with an opioid agonist medication (MAT+), those treated with an opioid antagonist medication (naltrexone) and OUD participants who are not being treated with medications (MAT-).

SECONDARY OUTCOMES:
1) To assess the impact of disruptions on striatal D1R to D2R availability on: DA release; Function of brain reward and control networks; Behavior.2) To assess if DA increases as achieved with oral MP influence the brain functional m... | End of study
  DA release (assessed with [11C]raclopride and the MP challenge strategy). Function of brain reward and control networks (assessed with fMRI with task activation and with RFC). Behavior (assessed with NP and actigraphy).
2) To assess if DA increases as achieved with oral MP influence the brain functional measures. | End of study
  Assess the association between striatal D1R to D2R availability and striatal DA release. Assess how D1R and D2R relate to behavior (locomotor activity and NP performance).
3) To assess if there is recovery after protracted treatment (comparing treated and non-treated) by repeating fMRI at 6 month follow-up. | End of study
  Determine if the brain recovers with protracted abstinence as assessed by recovery of resting brain networks and brain activation responses to stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Nora D Volkow Adler, M.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Data is analyzed by groups and not on an individual basis.

REFERENCES:
- [Derived] Zhang R, Manza P, Tomasi D, Kim SW, Shokri-Kojori E, Demiral SB, Kroll DS, Feldman DE, McPherson KL, Biesecker CL, Wang GJ, Volkow ND. Dopamine D1 and D2 receptors are distinctly associated with rest-activity rhythms and drug reward. J Clin Invest. 2021 Sep 15;131(18):e149722. doi: 10.1172/JCI149722. PMID 34264865
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-AA-0114.html